CLINICAL TRIAL: NCT06581601
Title: Physiotherapy Management in Women With Urinary Incontinence Considering Postural Stability, Postural Pattern, Pelvic Type, Quality of Life, and Sexual Aspect
Brief Title: Physiotherapy Management in Women With Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Małgorzata Wójcik, doctor, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2024
Record Dates: First submitted 2024-08-18; First posted 2024-09-03 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Urinary Incontinence
Keywords: the author's exercise program; urinary incontinence; physiotherapy
MeSH Terms: conditions — Urinary Incontinence | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Intervention Model Description: Pre- and post-menopause group perform author's exercise program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): 1.Contorl group: healtyhy women.
- Pre-menopausal group (Experimental): 2.Pre-menopasal group: experimental group - exercise's group
  Interventions: Other: physiotherapy, exercises
- Post-menopausal group (Experimental): 3.Post-menopausal group: experimental group - exercise's group
  Interventions: Other: physiotherapy, exercises

INTERVENTIONS:
Other: physiotherapy, exercises — An author's questionnaire will be used for participant selection, asking about the number and course of deliveries. Additionally, participants will log daily activities to calculate the physical activity level coefficient. Weight and height will be measured using a Tanita device to calculate BMI. The posture type and pelvic type will be assessed. Participants will be asked to complete the following questionnaires before and after the intervention: Pelvic Floor Disability Index (PFDI-20), Pelvic Floor Impact Questionnaire Short Form (PFIQ-7 SF), Sexual Satisfaction Scale (SSS-W-R15), Neck Disability Pain Index, Revised Oswestry Low Back Pain Disability Scale, Migraine Disability Assessment (MIDAS), Hospital Anxiety and Depression Scale (HADS), Short Form McGill Pain Questionnaire, CRANIA (Integrated Approach to Cranio Mandibular Neuroscience) questionnaire, IPAQ (International Physical Activity Questionnaire). Modified 1-Hour Pad Test. Execution of the Author's Training Program.
  Other Names: author's exercise program
  Arms: Post-menopausal group; Pre-menopausal group

SUMMARY:
Main objective:

The primary aim of the study is to assess whether the author's exercise programme has an effect on reducing urinary incontinence and pelvic floor dysfunction after childbirth, considering vacuum extractor, forceps and caesarean section deliveries.

Secondary objective:

The secondary objective is to determine whether the duration of the author's exercise programme is sufficient to achieve positive changes in women.

DETAILED DESCRIPTION:
The study will involve women with stress urinary incontinence, urge urinary incontinence, and mixed urinary incontinence. Participants will be women aged 20-80 years (meeting inclusion criteria: urinary incontinence, regular menstrual cycles, pre-and post menopausal period, natural childbirth or cesarean section, and deliveries using forceps and vacuum extractors; exclusion criteria: no urinary incontinence, irregular menstrual cycles, no childbirth, abdominal surgeries/procedures, active cancer, no gynecological check-up in the last 12 months, recurrent urogenital infections, joint hypermobility). A total of 300 women will be examined, including 100 women meeting the inclusion criteria, 100 women meeting the inclusion criteria but not interested in exercising, and 100 healthy women. Participants can withdraw from the study at any stage.Study Group Division

Based on the evaluation of posture type, pelvic pattern, and postural stability, participants will be divided into three groups:

1. Women meeting inclusion criteria performing the author's exercise program - experimental group.
2. Women meeting inclusion criteria but not interested in performing the author's exercise program - control group.
3. Healthy women - control group. The experimental group will perform the author's pelvic floor muscle exercise program daily for six weeks, at a fixed time each day, under weekly physiotherapist supervision and independently on other days (after proper instruction by the physiotherapist).

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence
* Regular menstrual cycles
* Pre and post-menopausal period
* Natural childbirth or cesarean section
* Deliveries using forceps and vacuum extractors

Exclusion Criteria:

* No urinary incontinence
* Irregular menstrual cycles
* No childbirth
* Abdominal surgeries/procedures Active cancer No gynecological check-up in the last 12 months Recurrent urogenital infections Joint hypermobility

Contorl group will be healthy women

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Modified 1-Hour Pad Test, measurement in grams | before start exercises and after six week finish exercises
  Before starting the author's six-week exercise program and after its completion, a modified 1-hour PAD Test will be conducted, which involves checking the amount of urine lost, during strictly defined activities. The test follows the guidelines in the literature. The test subject puts on a pre-weighed pad and, after emptying the bladder, drinks 500ml of water over 15 minutes. The test subject then waits 30 minutes. After this time, the test begins with 15 minutes of walking and climbing stairs. The test subject then performs a special training program: 10 times she stands up and sits down on a chair, 10 times she coughs vigorously, 10 times she picks up a bottle of water from the ground, runs in place for 1 minute, and for
  1 minute he holds his hands under running water. After the test is completed, the pad is weighed again and the amount of urine lost during the test is assessed.
Floor Disability Index | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Pelvic Floor Impact Questionnaire Short Form | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Sexual Satisfaction Scale | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Neck Disability Pain Index | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Revised Oswestry Low Back Pain Disability Scale | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Migraine Disability Assessment | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Hospital Anxiety and Depression Scale | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
Short Form McGill Pain Questionnaire | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
CRANIA (Integrated Approach to Cranio Mandibular Neuroscience) questionnaire | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The lower the value of the points received, the better the score.
International Physical Activity Questionnaire | before start exercises and after six week finish exercises
  Before the exercise begins and after it is completed, i.e. after 6 weeks, participants will fill out anonymously standardized questionnaires, in which they will have to mark the answer with an assigned score. The results will then be counted and scores will be assigned according to a key. The higher the value of the points received, the better the score.
Posture type Assessment by Hall-Wernham-Littlejohn, The result based on the observation of the posture with the use of the vertical, there is no measure or unit here. | before start exercises
  Type I correct: The examinee stands sideways, the plumb line is applied to the mastoid process of the temporal bone, correctly the plumb line runs along the cervical segment, through the middle of the shoulder, knee joint. For the front type II, the measurement is taken as before but the head is extended forward, the vertical course.Anterior pelvic tilt is still observed. With the rear type III, measurement as before. The vertical does not go through the center of the shoulder and knee. A posterior tilt of the pelvis, a rounded back and a receding head are observed.
Pelvic Type Assessment, result based on the evaluation of the height of the hip plates relative to the L4/L5 vertebra, there is no measure or unit here. | before start exercises
  The subject is standing and the examiner must identify the fourth and fifth lumbar vertebrae. Pelvic assessment is carried out according to Lewitt. Pelvis normal: If the iliac crests are at the height of the fourth and fifth lumbar vertebrae.The pelvis is highly assimilated when the iliac crests fall above the fourth and fifth lumbar vertebrae.Pelvic overload when the iliac crests fall below the fourth and fifth lumbar vertebrae.

SECONDARY OUTCOMES:
Postural stability assessment, measurement in the form of a number, the manufacturer does not provide measurement units. | before start exercises and after six week finish exercises
  Posturomed stablometric platform will be used to assess postural stability. Posturomed stablometric platform will be used to assess postural stability

CONTACTS AND LOCATIONS:
Overall Officials: Agata Wojtczak, Principal Investigator — Student Research Centre Conocimiento, Faculty of Sport Sciences in Gorzow Wielkopolski
Locations (1):
- 1Department of Physiotherapy, Poznan University of Physical Education, Faculty of Sport Sciences in Gorzow Wlkp., 61-871 Poznan, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
1. gathered groups.
  2. pre-exercise evaluation.
  3. exercises.
  4. post-exercise evaluation.
  5. Statistical compilation of data.
  6. Presentation of results at scientific conferences and in a scientific journal as a publication.